CLINICAL TRIAL: NCT06560281
Title: Effectiveness of Motion Minder Therapy (MoMT) Among Children With Spastic Hemiplegic Cerebral Palsy: A Pilot Study
Brief Title: Improving Hand Movements in Kids With One-Sided Arm Stiffness Cerebral Palsy Through Motion Minder Therapy (MoMT)
Acronym: MoMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Jeevarathinam Thirumalai, Principal Investigator, Saveetha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/032/2024/ISRB/SR/SCPT
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
Keywords: Cerebral Palsy; Spastic; Hemiplegic
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motion Minder Group (Experimental): Children in this arm receives a structured motion minder therapy protocol designed to improve fine motor skills in children with spastic hemiplegic cerebral palsy through targeted activities.
  Interventions: Other: Motion Minder Therapy (MoMT)

INTERVENTIONS:
Other: Motion Minder Therapy (MoMT) — Motion Minder Therapy (MoMT) total duration is 1 hour a day, 5 days a week for 4 weeks. The treatment is a carefully planned sequence of exercises intended to help children with spastic hemiplegic cerebral palsy develop their fine motor abilities. Activities includes Sticker Sorting, Beads on Parade, Pegboard Activities, Sensory Bins, Sculpture Building, Finger Painting & Drawing with Different Tools, Musical Instrument Play. Smartwatches that have tactile sensations and auditory indications are used strategically during certain tasks to enhance proprioception and give real-time feedback, making the rehabilitation process vibrant and interesting.

SUMMARY:
Motion Minder Therapy is a targeted intervention for fine motor skill challenges in spastic hemiplegic cerebral palsy children, emphasizing affordability, particularly in middle-income countries like India. Diverging from previous models requiring extensive daily supervision of 5 to 6 hours, Motion Minder Therapy optimizes resources by utilizing smartwatches for a focused 1-hour intervention. The study employs a Pilot phase with 5 children. Materials range from smart watch to sensory tools, offering a comprehensive approach. Statistical analysis, incorporating repeated measure ANOVA, aims to underscore Motion Minder Therapy's effectiveness in addressing the complex challenges of fine motor skill enhancement in spastic hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Beginning with a 5-minute Sticker Sorting exercise, the intervention aims to improve fine motor skills, hand-eye coordination, and cognitive abilities via the use of colorful stickers with varying sizes and textures. Children can then go on to the next activity during a quick 1-minute Rest & Reflection phase. In the eight-minute segment Beads on Parade, participants practice bilateral hand usage, fine motor coordination, and visual-motor integration by stringing colorful beads onto threads or wires. Pegboard Activities, an 8-minute exercise that emphasizes accuracy, hand strength, and spatial awareness through the positioning of pegs onto a board with corresponding holes, is preceded by another brief reflective pause. The following five-minute Sensory Bins practice promotes tactile exploration with objects like beans or rice, developing tactile sensitivity and sensory awareness. An eight-minute session called "Sculpture Building" focuses on developing hand strength, coordination, creativity, and fine motor abilities via the creation of three-dimensional shapes using clay. A 5-minute break is followed by Finger Painting & Drawing with Different Tools, an activity that uses a variety of painting tools to improve hand control and fine motor skills. The last part, a five-minute musical instrument play, comes after the last period of relaxation. Through tactile and aural experiences, children are encouraged to use hand to make various sounds and rhythms, encouraging bilateral coordination, fine motor control, and sensory integration.

ELIGIBILITY:
Inclusion Criteria:

* Age Eligibility: Children within the age bracket of 5 to 12 years.
* Manual Ability Classification System: Individuals falling into MACS categories I to III.
* Bimanual Fine Motor Function (BFMF): Participants falling within the BFMF spectrum of levels I to III.
* Modified Ashworth Scale (MAS): Participants falling within the MAS grade of I to III in upper extremity.
* Communication Functional Classification System (CFCS): Individuals with a CFCS classification ranging from I to III.
* Mini-Mental State Examination for Children: Individuals with Mini-Mental Examination score of 15.
* Grasping and Releasing Proficiency: Proficiency in grasping and releasing lightweight objects, with a minimum extension of 20° in the wrist and 10° in all Five metacarpophalangeal joints in the affected hand.

Exclusion Criteria:

* Presence of visual or auditory disorders.
* History of Seizure, respiratory issues and presence of hand deformities.
* Children who have undergone Botulinum neurotoxin injections or surgical interventions in the 6-month before study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Shriners Hospital Upper Extremity Evaluation (SHUEE) | Baseline, 4th week, 8th week, 12th week
  The Shriners Hospital Upper Extremity Evaluation is a video-based tool for the assessment of upper extremity function. The outcome is the total score of the spontaneous functional analysis, dynamic positional analysis, and grasp/release analysis. Total scores of 45 for spontaneous functional analysis, 72 for dynamic positional analysis and 6 for grasp/release. Higher scores mean a better outcome.
Nine Hole Peg Test | Baseline, 4th week, 8th week, 12th week
  Nine Hole Peg Test is used to measure the dexterity. Scores on nine-hole peg test are measured in seconds, indicating time taken to complete task. Higher scores indicate worse outcome, as they show slower completion times and reduced dexterity.

SECONDARY OUTCOMES:
Strengths and difficulties questionnaire | Baseline, 4th week, 8th week, 12th week
  The 25 item Strengths and Difficulties Questionnaire (SDQ) measures behavioral and emotional function. These 25 items are divided into 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The Strengths and Difficulties Questionnaire is scored on a 3-point Likert-type scale, with total scores (excluding the prosocial scale) ranging from 0 to 40. Higher scores reflect greater behavioral and emotional difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Prathap Suganthirababu, Ph.D.,, Study Chair — Saveetha University
Locations (2):
- India (2):
  - Saveetha Medical College and Hospital, Chennai, Tamil Nadu
  - Aadhuraa Special School, Kanchipuram, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn L, Ramasamy R, Dukes C, Scott J. Using WatchMinder to Increase the On-Task Behavior of Students with Autism Spectrum Disorder. J Autism Dev Disord. 2015 May;45(5):1408-18. doi: 10.1007/s10803-014-2300-x. PMID 25377769
- [Background] Jamali AR, Amini M. The Effects of Constraint-Induced Movement Therapy on Functions of Cerebral Palsy Children. Iran J Child Neurol. 2018 Fall;12(4):16-27. PMID 30279705
- [Background] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Background] Fong KN, Jim ES, Dong VA, Cheung HK. 'Remind to move': a pilot study on the effects of sensory cueing treatment on hemiplegic upper limb functions in children with unilateral cerebral palsy. Clin Rehabil. 2013 Jan;27(1):82-9. doi: 10.1177/0269215512448199. Epub 2012 Jul 16. PMID 22801471

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT06560281/Prot_SAP_ICF_002.pdf